CLINICAL TRIAL: NCT06017622
Title: Multi-center Observational Study of Plasma Concentrations of THC and Its Metabolites in Pediatric Patients Visiting Emergency Departments for Acute Cannabis-induced CNS Depression
Brief Title: Observational Study of THC Concentrations in Acute Cannabis-induced CNS Depression
Status: Active, not recruiting | Type: Observational
Sponsor: Anebulo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: AN01AC01
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Acute Cannabinoid Intoxication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for measurement of cannabinoid and metabolite concentrations in plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: There is a single group consisting of all subjects who meet the eligibility criteria

SUMMARY:
This observational study is being conducted to determine plasma concentrations of tetrahydrocannabinol (THC) and its metabolites, 11-OH-THC and THC-COOH, in plasma of subjects who visit the emergency department due to acute cannabinoid intoxication.

DETAILED DESCRIPTION:
This is a multi-center, prospective, cross-sectional observational study to determine the concentrations of tetrahydrocannabinol (THC) and its metabolites (and/or other cannabinoids) in the plasma of subjects admitted to emergency departments with acute cannabinoid intoxication The study will explore the relationships between these concentrations and parameters such as demographics, symptom severity, time to symptom resolution, and clinical outcomes.

Samples will be collected as part of standard clinical procedure without requiring study participants to spend additional time in the hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Subject visits emergency department for acute cannabinoid intoxication as evidenced by the following criteria:

   1. Recent cannabis use within the last 12 hours
   2. Clinically significant physiological abnormalities associated with cannabis use or problematic behavioral or psychological changes (e.g., altered perception, impaired motor coordination, euphoria, anxiety, a sensation of slowed time, impaired judgment, social withdrawal) that developed during, or shortly after, cannabis use
2. Subject (and/or parent/LAR when required) has the ability to communicate with comprehension with the study personnel at the time of consent/assent and the gathering of data other than plasma samples.
3. Subject (and/or parent/LAR when required) is willing and able to provide informed consent/assent.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

1. Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study.
2. Individuals under the age of 18 who do not have a parent or legal representative present during the time at the ED.
3. Patients presenting with signs or symptoms attributable to another medical condition or better explained by another mental disorder.
4. Patient presenting with cannabis hyperemesis syndrome (CHS) or cannabis withdrawal syndrome (CWS)
5. Patients who are brought in by law enforcement, i.e., cannabis intoxication associated with a vehicle accident (driving under the influence).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients of any age and sex who present to an emergency department with acute cannabinoid intoxication.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma Concentration of delta-9 tetrahydrocannabinol (THC) | Day 1
  Concentration of THC and THC metabolites (11-OH-THC and THC-COOH) in plasma of subjects admitted to emergency departments due to acute cannabinoid intoxication.

CONTACTS AND LOCATIONS:
Overall Officials: Ken Cundy, PhD, Study Director — Anebulo Pharmaceuticals Inc.
Locations (4):
- United States (4):
  - University of Colorado School of Medicine, Aurora, Colorado
  - Henry Ford Hospital, Detroit, Michigan
  - Oakland University William Beaumont School of Medicine, Royal Oak, Michigan
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No